CLINICAL TRIAL: NCT02821962
Title: Sedentary Intervention Trial in Cardiac Rehabilitation (SIT-CR): A Randomized Controlled Trial Using the activPAL3™ and activPAL3™ VT to Quantify Free-living Movement Patterns and Reducing Sedentary Time in Cardiac Rehabilitation Patients
Brief Title: Sedentary Intervention Trial in Cardiac Rehabilitation
Acronym: SIT-CR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ottawa Heart Institute Research Corporation (Other)
Collaborators: PAL Technologies Ltd. (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 20160336
Record Dates: First submitted 2016-06-17; First posted 2016-07-04 (Estimated); Results first posted 2019-06-10 (Actual); Last update posted 2019-07-17 (Actual); Status verified 2019-07

CONDITIONS: Coronary Artery Disease
Keywords: Sedentary behaviour
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Sedentary prompts (VTAP) (Experimental): Participants will complete supervised exercise sessions as part of cardiac rehabilitation programming on-site twice weekly for a total of 8 weeks. Participants will also be provided with a VTAP (activPAL3 VT) monitor to wear during waking hours for weeks 1 through 7 of cardiac rehabilitation. The VTAP will alert participants when they have been sedentary for 30 consecutive minutes.
  Interventions: Behavioral: Sedentary prompts from a VTAP device
- Usual care (No Intervention): Participants will complete supervised exercise sessions as part of cardiac rehabilitation programming on-site twice weekly for a total of 8 weeks.

INTERVENTIONS:
Behavioral: Sedentary prompts from a VTAP device
  Arms: Sedentary prompts (VTAP)

SUMMARY:
Exercise-based cardiac rehabilitation (CR) has been shown to consistently reduce the rates of total and cardiovascular-related mortality and morbidity. Sedentary behaviours have been shown to be high in patients with cardiovascular disease, but it is not yet known if current CR programming results in significant reductions in these behaviours, or whether a targeted component is warranted. It is also unclear if self-reported sedentary time measures can provide valid and reliable information for monitoring these behaviours in a CR setting, or whether more objective measures are needed. The purpose of this study is to assess the feasibility and usability of the activPAL3 devices for measuring sedentary time in a CR setting, describe changes in sedentary time that occur with standard CR and assess whether the addition of prompting cues from a device can result in further declines in sedentary behaviour and improvements in clinical outcomes, health related quality of life, symptoms of anxiety and depression, aortic stiffness, and aerobic capacity.

ELIGIBILITY:
Inclusion Criteria:

* Patient is attending on-site (2 times weekly for 8 weeks) cardiac rehabilitation at the Minto Prevention and Rehabilitation Centre at the University of Ottawa Heart Institute
* Patient is 18 years of age or older
* Patient has confirmed diagnosis of coronary artery disease (CAD)
* Patient understands English or French
* Patient is willing and able to provide informed consent

Exclusion Criteria:

* Patient is unwilling to wear activity monitors
* Patient is already using a commercial activity monitor with sedentary prompts (e.g. Jump Up, Garmin)
* Patient is unable to attend follow-up visits
* Patient not participating in a cardiac rehabilitation program at the University of Ottawa Heart Institute
* Patient has cognitive impairment (unable to comprehend or participate in the intervention)
* Patient has a history of postural hypotension
* Patient is unable, in the opinion of the Medical Director, to participate in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2016-08; Primary Completion 2017-09 (Actual); Study Completion 2017-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robert D Reid, PhD, MBA, Principal Investigator — Ottawa Heart Institute Research Corporation
Locations (1):
- University of Ottawa Heart Institute, Ottawa, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Sedentary Prompts (VTAP): Participants will complete supervised exercise sessions as part of cardiac rehabilitation programming on-site twice weekly for a total of 8 weeks. Participants will also be provided with a VTAP (activPAL3 VT) monitor to wear during waking hours for weeks 1 through 7 of cardiac rehabilitation. The VTAP will alert participants when they have been sedentary for 30 consecutive minutes.
  Sedentary prompts from a VTAP device
Period: Overall Study
Arm/Group | Sedentary Prompts (VTAP) | Usual Care
Started | 19 | 21
Completed | 17 | 21
Not Completed | 2 | 0
Not completed — Lost to Follow-up | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Sedentary Prompts (VTAP) | Usual Care | Total
Number analyzed (Participants) | 17 | 21 | 38
Age, Continuous [Mean (Standard Deviation); unit: years] | 62.4 (10.7) | 61.5 (9.7) | 61.9 (10.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 8 | 15
  Male | 10 | 13 | 23
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Count of Participants; unit: Participants]
  Canada | 17 | 21 | 38
Number of cardiac rehabilitation classes attended [Median (Inter-Quartile Range); unit: classes] | 14 [11 to 17] | 15 [13 to 17] | 14.5 [11.5 to 17]

OUTCOME MEASURES:

1. Primary Outcome: Feasibility and Usability of activPAL3 and VTAP Devices
Description: Primary objective is to assess the feasibility and usability of the activPAL3 and VTAP devices in a CR setting. Assessed by examining acceptability of intervention using evaluation surveys (scores). Reporting on number who reported willingness to wear the monitor again (3+). The scale is a 5-point Likert scale that asks "On a scale from 1 to 5, would you be willing to wear the monitor again?". Response options include: 1(never), 2, 3 (maybe), 4, and 5 (yes, please).
Time Frame: 9 weeks
Population: Those who completed and returned the satisfaction surveys.
Measure: Count of Participants; unit: Participants
Arm/Group | Sedentary Prompts (VTAP) | Usual Care
Number analyzed (Participants) | 14 | 19
Participants | 14 | 19

2. Secondary Outcome: Changes in Sedentary Time
Description: Changes in sedentary time measured by the activPAL3 over 8-week intervention period. Reported as proportion of day spent sedentary.
Time Frame: baseline and 8 weeks
Population: Those with complete baseline and post-intervention sedentary time (sitting + lying) measured via activPAL3
Measure: Mean (Standard Deviation); unit: Percentage of day
Arm/Group | Sedentary Prompts (VTAP) | Usual Care
Number analyzed (Participants) | 17 | 21
Percentage of day | -0.2 (10.6) | 1.9 (14.7)

3. Other Pre Specified Outcome: Changes in Moderate-to-vigorous Intensity Physical Activity
Description: Changes in moderate-to-vigorous intensity physical activity (measured by activPAL3)
Time Frame: baseline and 8 weeks
Population: Includes participants with complete data on moderate-to-vigorous intensity physical activity from baseline and 8 weeks.
Measure: Mean (Standard Deviation); unit: minutes/day
Arm/Group | Sedentary Prompts (VTAP) | Usual Care
Number analyzed (Participants) | 17 | 18
minutes/day | 10.62 (22.11) | 9.34 (15.95)

4. Other Pre Specified Outcome: Changes in Body Weight
Description: Changes in body weight (kg)
Time Frame: baseline and 8 weeks
Population: Includes participants with complete data on body weight from baseline and 8 weeks.
Measure: Mean (Standard Deviation); unit: kilograms
Arm/Group | Sedentary Prompts (VTAP) | Usual Care
Number analyzed (Participants) | 17 | 21
kilograms | -0.24 (2.64) | -0.08 (3.07)

5. Other Pre Specified Outcome: Changes in Clinical Body Mass Index
Description: Changes in body mass index (kg/m^2)
Time Frame: baseline and 8 weeks
Population: Includes participants with complete data on body mass index from baseline and 8 weeks.
Measure: Mean (Standard Deviation); unit: kilograms per meter squared
Arm/Group | Sedentary Prompts (VTAP) | Usual Care
Number analyzed (Participants) | 17 | 21
kilograms per meter squared | -0.07 (0.88) | -0.11 (1.14)

6. Other Pre Specified Outcome: Changes in Waist Circumference
Description: Changes in waist circumference (cm)
Time Frame: baseline and 8 weeks
Population: Includes participants with complete data on waist circumference from baseline and 8 weeks.
Measure: Mean (Standard Deviation); unit: centimeters
Arm/Group | Sedentary Prompts (VTAP) | Usual Care
Number analyzed (Participants) | 15 | 21
centimeters | -0.98 (3.98) | -4.45 (8.38)

7. Other Pre Specified Outcome: Changes in Systolic Blood Pressure
Description: Changes in systolic blood pressure (mmHg)
Time Frame: baseline and 8 weeks
Population: Includes participants with complete data on systolic blood pressure from baseline and 8 weeks.
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Sedentary Prompts (VTAP) | Usual Care
Number analyzed (Participants) | 17 | 21
mmHg | 1.65 (12.9) | 1.3 (14.7)

8. Other Pre Specified Outcome: Changes in Resting Heart Rate
Description: Changes in resting heart rate (bpm)
Time Frame: baseline and 8 weeks
Population: Includes those with complete data on resting heart rate at baseline and 8 weeks
Measure: Mean (Standard Deviation); unit: beats per minute
Arm/Group | Sedentary Prompts (VTAP) | Usual Care
Number analyzed (Participants) | 17 | 21
beats per minute | -1.3 (7.6) | -0.7 (8.2)

9. Other Pre Specified Outcome: Changes in Total Cholesterol
Description: Changes in total cholesterol (mmol/L)
Time Frame: baseline and 8 weeks
Population: Includes those with complete data on total cholesterol at baseline and 8 weeks
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Sedentary Prompts (VTAP) | Usual Care
Number analyzed (Participants) | 15 | 21
mmol/L | 0.05 (0.30) | 0.02 (0.69)

10. Other Pre Specified Outcome: Changes in HbA1c Percentage
Description: Changes in HbA1c percentage
Time Frame: baseline and 8 weeks
Population: Includes participants with complete data on HbA1c % from baseline and 8 weeks.
Measure: Mean (Standard Deviation); unit: percentage
Arm/Group | Sedentary Prompts (VTAP) | Usual Care
Number analyzed (Participants) | 14 | 21
percentage | -0.01 (0.27) | 0.26 (0.73)

11. Other Pre Specified Outcome: Changes in Anxiety
Description: Changes in measures of anxiety as assessed using the Hospital Anxiety and Depression Scale. Lower scores mean a better outcome. Score ranges from 0 to 21.
Time Frame: baseline and 8 weeks
Population: Includes participants with complete data on anxiety from the HADS from baseline and 8 weeks.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Sedentary Prompts (VTAP) | Usual Care
Number analyzed (Participants) | 13 | 17
score on a scale | -1.7 (2.5) | -3.1 (3.7)

12. Other Pre Specified Outcome: Changes in Health-related Quality of Life (Physical Component Scale)
Description: Changes in health-related quality of life (Physical Component Scale) as measured by the Short Form-36. Higher scores represent better physical health. Range 0 -100
Time Frame: baseline and 8 weeks
Population: Includes participants with complete data on quality of life from baseline and 8 weeks.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Sedentary Prompts (VTAP) | Usual Care
Number analyzed (Participants) | 16 | 21
score on a scale | 6.9 (3.8) | 3.2 (4.7)

13. Other Pre Specified Outcome: Changes in Pulse Wave Velocity
Description: Changes in pulse wave velocity
Time Frame: baseline and 8 weeks
Population: Includes participants with complete data on pulse wave velocity from baseline and 8 weeks.
Measure: Mean (Standard Deviation); unit: m/s
Arm/Group | Sedentary Prompts (VTAP) | Usual Care
Number analyzed (Participants) | 16 | 21
m/s | 0.01 (0.34) | 0.10 (0.42)

14. Other Pre Specified Outcome: Changes in Maximal Aerobic Power (VO2peak)
Description: Changes in maximal aerobic power as assessed using a Modified Bruce Ramp Treadmill Test
Time Frame: baseline and 8 weeks
Population: Includes participants with complete data on VO2 peak from baseline and 8 weeks.
Measure: Mean (Standard Deviation); unit: mL/kg/min
Arm/Group | Sedentary Prompts (VTAP) | Usual Care
Number analyzed (Participants) | 17 | 21
mL/kg/min | 1.62 (6.09) | 1.70 (4.50)

15. Other Pre Specified Outcome: Change in Health-related Quality of Life (Mental Component Scale)
Description: Change in health-related quality of life (Mental Component Scale) from the SF-36. Higher scores represent better mental health. Range 0 to 100.
Time Frame: baseline and 8 weeks
Population: Includes participants with complete data on health-related quality of life from baseline and 8 weeks.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Sedentary Prompts (VTAP) | Usual Care
Number analyzed (Participants) | 16 | 21
score on a scale | 1.8 (10.7) | 2.7 (7.1)

16. Other Pre Specified Outcome: Changes in HDL
Description: Changes in HDL
Time Frame: baseline and 8 weeks
Population: Includes participants with complete data on HDL from baseline and 8 weeks.
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Sedentary Prompts (VTAP) | Usual Care
Number analyzed (Participants) | 15 | 21
mmol/L | 0.12 (0.15) | 0.09 (0.12)

17. Other Pre Specified Outcome: Changes in Depression Symptoms as Measured by the Hospital Anxiety and Depression Scale.
Description: Changes in depression symptom score. Lower scores mean a better outcome. Score ranges from 0 to 21.
Time Frame: baseline and 8 weeks
Population: Includes participants with complete data on depression scores from baseline and 8 weeks.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Sedentary Prompts (VTAP) | Usual Care
Number analyzed (Participants) | 11 | 19
score on a scale | -0.7 (2.6) | -1.8 (4.2)

ADVERSE EVENTS:
Time Frame: 9 weeks
Arm/Group | Sedentary Prompts (VTAP) | Usual Care
All-Cause Mortality (participants affected / at risk) | 0/19 | 0/21
Serious Adverse Events (participants affected / at risk) | 0/19 | 0/21
Other Adverse Events (participants affected / at risk) | 0/19 | 0/21

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-07-25): https://cdn.clinicaltrials.gov/large-docs/62/NCT02821962/Prot_SAP_000.pdf